CLINICAL TRIAL: NCT07193953
Title: Targeting Neuroinflammation With Enhanced Delivery of Intravenous Immunoglobulin to the Motor Cortex Using Next Generation Dome Helmet Focused Ultrasound in Amyotrophic Lateral Sclerosis: A Phase I, Open Label Trial
Brief Title: Intravenous Immunoglobulin (IVIG) and Blood-Brain Barrier Disruption in Amyotrophic Lateral Sclerosis (ALS)
Acronym: ALSFUS003
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Principal Investigator, Dr. Nir Lipsman, Chief of Hurvitz Brain Sciences Program, Director of Harquail Centre for Neuromodulation, Director of Neurosurgery Residency Program, Principal Investigator, Associate Professor, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 6271
Record Dates: First submitted 2025-05-12; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: ALS; Focused Ultrasound; Blood Brain Barrier Opening; Intravenous Immunoglobulin; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Immunoglobulins, Intravenous; Solutions

STUDY DESIGN:
Intervention Model Description: The first cohort (n = 3) will receive 0.4g/kg of IVIg, divided into two 0.2g/kg doses. After a preliminary safety and tolerability assessment of the first cohort, patients will be enrolled to the second cohort (n = 3). It will follow the same design but with 0.8g/kg divided into two 0.4g/kg doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous Immunoglobulin Administration using Focused Ultrasound (Experimental): ALS patients will be assigned to receive Intravenous Immunoglobulin (IVIg) and DEFINITY® microbubbles. The first three enrolled patients will participate in the first cohort, receiving 0.4g/kg divided in two doses. After a preliminary safety assessment of the first cohort, the next three successfully screened patients will be enrolled in the second cohort, receiving 0.8g/kg divided in two doses. The second IVIg dose in each cohort will be administered in combination with Next Generation Dome Helmet (NGDH) focused ultrasound (FUS) to transiently open the blood-brain barrier and enhance IVIg delivery to the primary motor cortex.
  Interventions: Device: Next Generation Dome Helmet Focused Ultrasound; Drug: Intravenous immunoglobulin (IVIG), 10% solution for infusion; Drug: Definity® Vial for (Perflutren Lipid Microsphere) Injectable Suspension

INTERVENTIONS:
Device: Next Generation Dome Helmet Focused Ultrasound — Two doses of IVIg will be administered 2 weeks apart. The first dose at Week 0 will be a standalone administration. The second dose at Week 2 will be combined with Next Generation Dome Helmet (NGDH) Focused Ultrasound (FUS) blood brain barrier (BBB) opening.
Drug: Intravenous immunoglobulin (IVIG), 10% solution for infusion — Two doses of IVIg will be administered 2 weeks apart. The first dose at Week 0 will be a standalone administration. The second dose at Week 2 will be combined with Next Generation Dome Helmet (NGDH) Focused Ultrasound (FUS) blood brain barrier (BBB) opening. Cohort I will receive 0.2g/kg of IVIg at each dose. Cohort II will receive 0.4g/kg of IVIg at each dose.
  Privigen® IVIg comes in vials containing 10% active ingredient. It is supplied in 2.5 g (25 mL bottle), 5 g (50 mL bottle), 10 g (100 mL bottle), 20 g (200 mL bottle) or 40 g (400 mL bottle). The IVIg dose will be determined based on the patient's ideal body weight.
Drug: Definity® Vial for (Perflutren Lipid Microsphere) Injectable Suspension — DEFINITY® Perflutren Injectable Microbubbles is an ultrasound contrast imaging agent that will be used for blood brain barrier opening during focused ultrasound. These microbubbles will be injected during the focused ultrasound procedure on the day of the second IVIg dose.

SUMMARY:
The goal of this study is to evaluate the safety and feasibility of IVIg administration in conjunction with primary motor cortex BBB opening using the Next Generation Dome Helmet (NGDH) FUS in adult participants with ALS.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label, multiple-ascending dose (MAD), phase I trial to evaluate safety, feasibility, pharmacodynamics, and pharmacokinetics of enhanced delivery of IVIg 0.4 or 0.8g/kg to the primary motor cortex in 6 patients with ALS by using a single BBB opening procedure targeting the primary motor cortex in both brain hemispheres. Six participants will be enrolled in two sequential cohorts. The first cohort (n = 3) will receive 0.4g/kg of IVIg divided in two doses, while the second cohort (n = 3) will receive a 0.8g/kg of IVIg divided in two doses. In both cohorts, the second dose of IVIg will be accompanied by a single BBB opening procedure targeting the primary motor cortex in both brain hemispheres with focused ultrasound (FUS) using Next Generation Dome Helmet and intravenous microbubbles (DEFINITY®, Lantheus Medical Imaging Canada, Inc., Montreal, QC, Canada). This FUS procedure will occur during 2 weeks after the first dose administration. Follow-up visits will occur over the span of 24 weeks from the first dose.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with ALS as per the Gold Coast Criteria;
2. Aged 18 years or older;
3. Capable of providing informed consent and complying with study procedures;
4. If taking Riluzole, on a stable dose for at least 4 weeks prior to Baseline;
5. If taking Edaravone, on a stable dose of one completed cycle prior to Baseline;
6. Respiratory Function Criterion:

   * Able to lie supine without BiPAP or breathing discomfort; OR
   * Forced vital capacity or slow vital capacity ≥50% of the predicted value for sex, height and age, if available
7. Able to communicate sensations during the Dome FUS procedure.
8. Qualified fit for the anesthesia by an anesthesiologist, ASA I-III.

Exclusion Criteria:

1. MRI findings:

   1. Active infection/inflammation
   2. Acute or chronic hemorrhages, specifically > 4 lobar microbleeds, and no siderosis or macrohemorrhages
   3. Tumor/space occupying lesion causing significant mass effect
   4. Meningeal enhancement
   5. Intracranial hypotension
2. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
3. Clips or other metallic implanted objects in the skull or the brain, except shunts
4. Significant cardiac disease or unstable hemodynamic status including:

   1. Documented myocardial infarction within six months of screening
   2. Unstable angina on medication
   3. Unstable or worsening congestive heart failure
   4. Left ventricular ejection fraction below the lower limit of normal
   5. History of a hemodynamically unstable cardiac arrhythmia
   6. Cardiac pacemaker
   7. Severe hypertension (diastolic BP > 100 on medication)
   8. Patient has right-to-left, bidirectional, or transient right-to-left cardiac shunts
   9. QT prolongation observed on screening ECG (QTc > 450 for men and > 470 for women)
5. Uncontrolled hypertension (systolic > 150 and diastolic BP > 100 on medication)
6. Patients should not take medications known to increase risk of hemorrhage (e.g., aspirin or class I and III anticoagulants) for at least 7 days prior to treatment or lumbar puncture; patients should not take Avastin for 30 days prior to treatment
7. History of a bleeding disorder, coagulopathy or a history of spontaneous hemorrhage or use of anticoagulants, specifically recent thrombosis or stroke in past 3 months; abnormal coagulation profile (PLT < 100,00/μl), PT (> 14 sec) or PTT (> 36 sec), and INR > 1.3
8. No more than 1 non-strategic lacune <1.5 cm
9. Known cerebral or systemic vasculopathy
10. Significant depression and at potential risk of suicide
11. Known sensitivity/allergy to gadolinium (an alternative product may be used) and DEFINITY®.
12. Any contraindications to MRI scanning, including:

    1. Large participants not fitting comfortably into the scanner
    2. Difficulty lying supine and still for up to 3 hours in the MRI unit or claustrophobia
13. Any contraindication to lumbar puncture for collection of cerebral spinal fluid, including:

    a. Intracranial hypotension
14. Untreated, uncontrolled sleep apnea
15. Impaired renal function with estimated glomerular filtration rate < 30 mL/min/1.73m2 or on dialysis.
16. IVIg use in the previous 6 months.
17. Live viral vaccination within the 30 days before study entry
18. Currently, or in the last 3 months participated in a clinical trial delivering an investigational product or non-approved use of a drug or device or in any other type of medical research.
19. Respiratory: chronic pulmonary disorders e.g. severe emphysema, pulmonary vasculitis, or other causes of reduced pulmonary vascular cross-sectional area, patients with a history of drug allergies, uncontrolled asthma or hay fever, and multiple allergies where the benefit/risk of administering DEFINITY® is considered unfavorable by the study physicians in relation to the product monograph for DEFINITY®.
20. Motor cortex atrophy deemed severe enough to limit targeting
21. Previous major allergic or anaphylactic reaction to IVIg
22. Known IgA deficiency with anti-IgA.
23. Known frontotemporal dementia;
24. Definitely or possibly pregnant (if applicable);
25. Known auto-immune condition with or without neurological manifestations (e.g., multiple sclerosis (MS), systemic lupus erythematous (SLE), Rheumatoid arthritis).
26. Current, planned or previous use of oral, intramuscular or intravenous steroid drugs (such as prednisone, prednisolone, dexamethasone, triamcinolone, methylprednisolone, oxandrolone, and others), immunosuppressant drugs (azathioprine, mycophenolate, tacrolimus, sirolimus, cyclophosphamide, and others) or NSAIDs (ibuprofen, naproxen, celecoxib, and others) in the past 30 days;
27. Other unspecified reasons that, in the opinion of the Investigator or the Sponsor, make the participant unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Safety of IVIg in patients with ALS | During and after IVIg administration at Week 0 and Week 2 Day 1 until Week 24.
  This will be assessed up through the incidence of drug-related adverse events, serious adverse events, and discontinuations due to adverse events after Intravenous Immunoglobulin (IVIg) administration.
Safety of DEFINITY® microbubbles | During and after DEFINITY® administration at Week 2 Day 1 until Week 24.
  This will be assessed up through the incidence of drug-related adverse events, serious adverse events, and discontinuations due to adverse events after DEFINITY® infusion during focused ultrasound (FUS) blood brain barrier (BBB) opening.
Feasibility of FUS BBB opening in the motor cortex | During and after Week 2 Day 1 FUS BBB opening until Week 24.
  This will be measured as detectable gadolinium enhancement at the arm, leg and bulbar regions of the motor cortex bilaterally following FUS with posterior normalization.
Safety of FUS BBB opening in the motor cortex | From up to 30 days before Week 0 to Week 24.
  Incidence of BBB opening-related and FUS-related adverse events, serious adverse events, incidence of asymptomatic or symptomatic radiologic complication, such as evidence of bleeding or swelling after FUS, incidence of electrographic complication, such as epileptiform discharges on EEG, or accelerated ALS disease progression, defined as ≥ 6-point decline in the ALSFRS-R scores from Baseline to week 8.

SECONDARY OUTCOMES:
Neurofilament light chain (NfL) levels in blood plasma and cerebrospinal fluid | From up to 30 days before Week 0 to Week 24.
  Change in concentration of serum neurofilaments from Baseline to Week 24
Inflammatory markers in blood and cerebrospinal fluid | From up to 30 days before Week 0 to Week 24.
  Change in cerebrospinal fluid (CSF) and blood inflammatory markers, including but not limited to TNF-α, IL-1β, IL-2, IL-6, IL-8, IL-17, CHIT1, CHI3L1, CHI3L2, TGF-β, IL-10, and CRP

OTHER OUTCOMES:
Pharmacokinetics Outcome - Immunoglobulin G Concentration | From up to 30 days before Week 0 to Week 24.
  Change in the cerebrospinal fluid (CSF)/whole blood ratio of Immunoglobulin G (IgG) concentration. This will serve as a pharmacokinetics outcome of enhanced IVIg delivery to the central nervous system after blood brain barrier opening.
Exploratory Outcomes - ALSFRS-R scores | From up to 30 days before Week 0 to Week 24.
  A ≥ 4-point increase in the Amyotrophic Lateral Sclerosis Functional Rating Scale Revised (ALSFRS-R) scores or significant clinical improvement at week 8.
Exploratory Outcomes - Changes in levels of cerebral chemicals measured using Magnetic Resonance Spectroscopy | From up to 30 days before Week 0 to Week 24.
  Changes in cerebral chemicals through Magnetic Resonance Spectroscopy (MRS). These include N-acetylaspartate (NAA), total choline (Cho), total creatine (Cr), myo-inositol (Ino), Glutamate (Glu), and Gamma-aminobutyric acid (GABA). All measurements use the same units.
Pharmacokinetics Outcome - Neurofilament light chain levels | From up to 30 days before Week 0 to Week 24.
  Change in cerebrospinal fluid and blood neurofilament light chain (NfL) post Next Generation Dome Helmet Focused Ultrasound (FUS) procedure, from week 2 to 24. This will serve as a pharmacokinetic outcome of NfL behavior post FUS procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No